CLINICAL TRIAL: NCT00333554
Title: Nutritional Intervention to Prevent Diabetes
Acronym: TN06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TN06 NIP; UC4DK097835 (NIH)
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: DHA; docosahexaenoic acid; omega-3 fatty acid; fish oil; pregnancy; infancy; prevention; "at risk" for developing type 1 diabetes; juvenile diabetes; T1D; diabetes mellitus; Type 1 diabetes TrialNet; TrialNet; dietary supplementation; nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA Treatment Group (Experimental): DHA study treatment given on daily basis to nursing mother (breast milk) or baby as either formula, or capsules (removing content and mixing with food)depending on age of child.
  Interventions: Dietary Supplement: DHA Treatment
- Control Group (Placebo Comparator): Placebo for DHA given to nursing mother (breast milk), study formula, or capsules (removing content and mixing with food)depending on age of child.
  Interventions: Dietary Supplement: Placebo for DHA

INTERVENTIONS:
Dietary Supplement: DHA Treatment — DHA study treatment given on daily basis to nursing mother (breast milk) or baby as either formula, or capsules (removing content and mixing with food) depending on age of child.
  Arms: DHA Treatment Group
Dietary Supplement: Placebo for DHA — Study placebo given on daily basis to nursing mother (breast milk) or baby as either formula, or capsules (removing content and mixing with food)depending on age of child.
  Arms: Control Group

SUMMARY:
Type 1 Diabetes (T1D) is an autoimmune disease. This means that the immune system (the part of the body which helps fight infections) mistakenly attacks and destroys the cells that produce insulin (islet cells found in the pancreas). As these cells are destroyed, the body's ability to produce insulin decreases.

The autoimmune process is thought to be initiated by a gene-environment interaction. The genetics involved in the development of T1D are fairly well understood. There is a higher risk of developing T1D with the presence of the human leukocyte antigen (HLA) DR3 or DR4. It is also known that not everyone with these genes actually develops T1D. Therefore, one or more environmental factors are thought to contribute to the process of developing T1D.

The consumption of the anti-inflammatory fatty acids, the omega-3 fatty acids, has decreased significantly in the past 100 years. At the same time a rise in the incidence of T1D, especially in young children has occurred. Because of the warnings to eliminate fish during pregnancy, pregnant women are consuming even less omega-3 fatty acids during fetal development.

Observations have been made that children who have received omega-3 fatty acid supplementation have a lower risk of T1D. Omega-3 fatty acids could have a protective effect that may occur during pregnancy, infancy, or both. The mechanism of this protection may be due to the DHA mediated suppression of the inflammatory response.

Patients at higher risk for T1D have an increased pro-inflammatory environment. We hypothesize that DHA supplementation during pregnancy and early childhood will block the initial pro-inflammatory events and prevent development of islet cell autoimmunity in children at higher risk for T1D.

This study is a feasibility study to determine if a full-scale DHA supplementation study will be implemented. If a full study is implemented, the primary outcome will be to determine if nutritional supplementation with omega-3 fatty acids during the last trimester of a mother's pregnancy and/or the first three years of life for children who are at higher risk of T1D will prevent the development of islet autoimmunity.

DETAILED DESCRIPTION:
There are two possible entry pathways for study participants. The first pathway is the entry point for pregnant mothers in their third trimester (24 weeks gestational age) whose babies may be at higher risk for T1D based on family history. At birth, or soon after, their babies will be tested for HLA type (to look for the specific gene which confers a higher risk of developing T1D). If the HLA typing shows that the baby is at higher risk for T1D and no protective genes are present, the baby will then continue in the study. The second pathway is the entry point for babies whose mothers were not enrolled during pregnancy. These babies will also be tested for HLA type. Their eligibility will be based on the presence of higher risk genes or the presence of a multiplex family history. This screening process may take place up until the baby is 5 months old.

Eligible participants (pregnant women or infants) will be randomized to one of the two study groups: DHA (docosahexaenoic acid) study substance (this is the intervention) or control study substance (this is the placebo). The DHA (docosahexaenoic acid) to be used in this trial is produced from algae, not from fish oil, so there is no risk of mercury or pesticide contamination.

Pregnant and nursing mothers who are assigned to the control group will receive study capsules containing a vegetable oil and no DHA (docosahexaenoic acid) . Pregnant and nursing mothers who are assigned to the experimental group will receive study capsules containing DHA (docosahexaenoic acid) . During pregnancy and while breastfeeding, infants will receive the study substance indirectly through their mother (either the placenta or breastmilk).

Infants who are either partially or exclusively formula feeding will receive study substance more directly through the study formula. The control group will receive study formula containing the typical amount of DHA that can be found in some infant formulas, while infants in the experimental group will receive study formula containing a larger amount of DHA (docosahexaenoic acid) than typically found in some infant formulas. By six to twelve months of age, all infants will get study supplement added to solid foods.

All mothers will have contact with the study site every 3 months. Nursing mothers will provide samples of breast milk for fatty acids analysis at these visits.

Infants will need to come to follow-up study visits every 6 months. At each of these visits, the infant will have a limited physical exam and blood drawn from a vein to monitor immune activity, levels of fatty acid and vitamin D, and to check for diabetes-related autoantibodies. Infants/children cannot continue in the study if they: (1) develop two positive autoantibodies, present at two consecutive visits, or (2) develop T1D.

All follow-up study visits will continue for 1-2 years, and possibly an additional 2 years if a full-scale study is initiated.

ELIGIBILITY:
Inclusion Criteria

Pregnant mothers are eligible for enrollment into this study if they:

1. Have T1D or the child's father, or a full or half-sibling of the child has T1D
2. Are 18 years of age or older
3. Are in their third trimester of pregnancy (i.e. gestation is 24 weeks or longer)
4. Have understood and signed a written informed consent and HIPAA authorization
5. Are willing to undergo randomization to ensure that equal numbers receive the DHA study substance versus the control

Infants are eligible for enrollment into this study if they:

1. Are less than or equal to six months of age on the date of randomization
2. Are found to be at risk for type 1 diabetes because they have a mother, father or full or half-sibling with T1D AND

   * have a DR3 or DR4 allele OR
   * have another relative (includes both 1st and 2nd degree relatives) with T1D (multiplex family)
3. Have a parent or legal guardian who has understood and signed a written informed consent and HIPAA authorization
4. Have a parent(s) or legal guardian(s) who are willing for their baby to undergo randomization to ensure that equal numbers receive the DHA study substance versus the control

Exclusion Criteria

Pregnant mothers are NOT eligible for enrollment into this study if they:

1. Have any condition the investigator believes will put the mother or her fetus at an unacceptable medical risk for participation in this study
2. Have a known complication of pregnancy causing an increased risk for the mother or fetus prior to entry into the study
3. Have previously had multiple (2 or more) pre-term births (<36 weeks)
4. Are diabetic and have a known HbA1c greater than 9% at anytime during the pregnancy (however, healthy infants after birth may qualify in spite of the above restrictions during pregnancy)
5. Plan to take DHA supplementation during the study

Infants are NOT eligible for enrollment into this study if they:

1. Have any condition the investigator believes will put the subject at an unacceptable medical risk for participation in this study
2. Have a mother with a condition the investigator believes will put her at an unacceptable medical risk for participation in this study
3. Have a nursing mother who plans to take DHA supplementation or has a parent or legal guardian who plans to provide supplementation to his/her infant independently during the study
4. Have a protective allele (DQB1*0602 or DRB1*0403)
5. Were born prior to 36 weeks gestation and require a pre-term infant formula

Max Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
20% higher level of plasma and/or red blood cell membrane phospholipid DHA achieved in the treatment group | Every 3 months for two years; every 6 months until age 3.
At least a 20% reduction in the level of the major inflammatory cytokine, IL1-beta, achieved in the plasma of the treatment group | Every 3 months for two years; every 6 months until age 3.

SECONDARY OUTCOMES:
95% of families will continue to attend follow-up visits | Every 3 months for two years; every 6 months until age 3.

CONTACTS AND LOCATIONS:
Overall Officials: Jay S Skyler, M.D., Study Chair — University of Miami; H. Peter Chase, MD, Principal Investigator — The University of Colorado Health Science Center- Barbara Davis Center for Childhood Diabetes; Michael Clare-Salzler, MD, Principal Investigator — University of Florida, Department of Pathology, Department of Pediatrics, Diabetes Research Program
Locations (9):
- United States (9):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, San Francisco, San Francisco, California
  - Indiana University-Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Health Care, Iowa City, Iowa
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Utah Diabetes Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/tn06-nip-pilot/?query=tn06
URL: https://repository.niddk.nih.gov/studies/tn06-nip-pilot/?query=tn06

REFERENCES:
- [Background] Verge CF, Gianani R, Kawasaki E, Yu L, Pietropaolo M, Jackson RA, Chase HP, Eisenbarth GS. Prediction of type I diabetes in first-degree relatives using a combination of insulin, GAD, and ICA512bdc/IA-2 autoantibodies. Diabetes. 1996 Jul;45(7):926-33. doi: 10.2337/diab.45.7.926. PMID 8666144
- [Background] Karvonen M, Pitkaniemi J, Tuomilehto J. The onset age of type 1 diabetes in Finnish children has become younger. The Finnish Childhood Diabetes Registry Group. Diabetes Care. 1999 Jul;22(7):1066-70. doi: 10.2337/diacare.22.7.1066. PMID 10388969
- [Background] Rice R. Fish and healthy pregnancy: more than just a red herring! Prof Care Mother Child. 1996;6(6):171-3. PMID 9077255
- [Background] Stene LC, Joner G; Norwegian Childhood Diabetes Study Group. Use of cod liver oil during the first year of life is associated with lower risk of childhood-onset type 1 diabetes: a large, population-based, case-control study. Am J Clin Nutr. 2003 Dec;78(6):1128-34. doi: 10.1093/ajcn/78.6.1128. PMID 14668274
- [Background] Endres S, Ghorbani R, Kelley VE, Georgilis K, Lonnemann G, van der Meer JW, Cannon JG, Rogers TS, Klempner MS, Weber PC, et al. The effect of dietary supplementation with n-3 polyunsaturated fatty acids on the synthesis of interleukin-1 and tumor necrosis factor by mononuclear cells. N Engl J Med. 1989 Feb 2;320(5):265-71. doi: 10.1056/NEJM198902023200501. PMID 2783477
- [Background] Simopoulos AP. Essential fatty acids in health and chronic disease. Am J Clin Nutr. 1999 Sep;70(3 Suppl):560S-569S. doi: 10.1093/ajcn/70.3.560s. PMID 10479232
- [Background] Chase HP, Cooper S, Osberg I, Stene LC, Barriga K, Norris J, Eisenbarth GS, Rewers M. Elevated C-reactive protein levels in the development of type 1 diabetes. Diabetes. 2004 Oct;53(10):2569-73. doi: 10.2337/diabetes.53.10.2569. PMID 15448085
- [Background] Friedberg CE, Janssen MJ, Heine RJ, Grobbee DE. Fish oil and glycemic control in diabetes. A meta-analysis. Diabetes Care. 1998 Apr;21(4):494-500. doi: 10.2337/diacare.21.4.494. PMID 9571330
- [Result] Chase HP, Boulware D, Rodriguez H, Donaldson D, Chritton S, Rafkin-Mervis L, Krischer J, Skyler JS, Clare-Salzler M; Type 1 Diabetes TrialNet Nutritional Intervention to Prevent (NIP) Type 1 Diabetes Study Group. Effect of docosahexaenoic acid supplementation on inflammatory cytokine levels in infants at high genetic risk for type 1 diabetes. Pediatr Diabetes. 2015 Jun;16(4):271-9. doi: 10.1111/pedi.12170. Epub 2014 Jul 12. PMID 25039804
- See also: Related Info — http://www.diabetestrialnet.org/
- See also: Related Info — http://www.jdrf.org/